CLINICAL TRIAL: NCT07205575
Title: AI-Guided Proteomic Discovery and Multi-Cohort Validation of a Circulative Protein Signature to Differentiate Bacterial and Viral Infections in Acute Febrile Illness
Brief Title: AI-Guided Proteomic Biomarker Panel for Differentiating Bacterial and Viral Infections in Acute Febrile Illness
Status: Completed | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Gang Wang, MD, Principal Investigator, Qilu Hospital of Shandong University
Other Study IDs: KYLL-202008-058-P; 2021SDUCRCC004 (Other: Ethics Committee of Shandong University of Qilu Hospital)
Record Dates: First submitted 2025-09-15; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Acute Febrile Illness; Bacterial Infections; Viral Infections; Sepsis
MeSH Terms: conditions — Bacterial Infections; Virus Diseases; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bacterial infections: Individuals with acute fever whose positive bacteria isolated from sterile or non-sterile sites have pathological characteristics.
  Interventions: Diagnostic Test: Proteomic Biomarker Panel
- Viral infections: Group/Cohort Description: Individuals with acute fever whose viral nucleic acid test and/or serological positive compatible with acute syndrome#(e.g. serology, PCR).
  Interventions: Diagnostic Test: Proteomic Biomarker Panel

INTERVENTIONS:
Diagnostic Test: Proteomic Biomarker Panel — A blood-based ELISA test measuring circulating ICAM1, CFHR5, and GRN. Index test performance will be evaluated against microbiological gold standards and adjudication.

SUMMARY:
This study is a proteomics-based diagnostic biomarker study conducted on the same patient cohort as the transcriptomic biomarker study (NCT065529754). Although both studies share the same clinical cohort and overarching diagnostic aim, they are registered separately because they employ distinct omics technologies, investigate different biomarker modalities, and yield independent outcome measures.

DETAILED DESCRIPTION:
This study aims to identify and validate proteomics-based diagnostic biomarkers for differentiating bacterial from viral acute febrile illnesses. It is conducted on the same patient cohort previously used in a registered transcriptomic biomarker study (ClinicalTrials.gov Identifier: NCT065529754).

Although both studies share the overarching clinical objective of improving infection triage, they are scientifically independent in terms of methodology, biomarker modality, and analytical pipeline. Transcriptomic study (NCT065529754): Focused on host-response gene expression signatures derived from RNA sequencing data. Proteomic study (this registration): Focuses on host-response protein biomarkers identified through high-resolution mass spectrometry (DIA/PRM/SRM) and validated by immunoassays (ELISA).

The proteomics study is designed to discover a minimal and biologically distinct set of protein markers that can be readily translated into clinical diagnostics. This study evaluates a minimal set of circulating proteins-ICAM1, CFHR5, and GRN-discovered through AI-assisted proteomics and validated by ELISA, as a rapid diagnostic tool for bacterial vs viral infection. Patients with acute fever are prospectively enrolled into three cohorts: discovery, internal validation, and external validation.

This independent registration reflects the proteomics-specific objectives, methodology, and outcomes, while also acknowledging its linkage to the transcriptomics study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥14 years；
* Body temperature > 38°C(within the past 72 hours)；
* Disease duration ≤ 14 days；
* Provision of informed consent by patient or legal guardian.

Exclusion Criteria:

* Underlying diseases affecting immune function (e.g., advanced malignancy, autoimmune disease, immunodeficiency, use of immunosuppressants);
* Pregnancy;
* Mixed infections (including viral-bacterial co-infections, bacterial or viral-fungal co-infections, or autoimmune disease concomitant with bacterial infection);
* indeterminate or negative microbiological testing ;
* inability to provide informed consent

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 14 years or older who presented to the emergency department with acute febrile illness (fever ≤14 days, ≥38°C within 72 hours) and suspected bacterial or viral infection.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy (AUROC) for differentiating bacterial vs viral infection | At hospital admission (retrospective review of cases from September 1, 2021 to October 31, 2024)
  The area under the receiver operating characteristic curve (AUROC) will be calculated for the selected host-response protein biomarker panel to assess its ability to discriminate bacterial from viral infections in patients presenting with acute febrile illness.

SECONDARY OUTCOMES:
Incremental diagnostic value of biomarker panel combined with CRP | At hospital admission (retrospective review of cases from September 1, 2021 to October 31, 2024)
  Evaluate the increase in area under the receiver operating characteristic curve (AUROC) when the host-response protein biomarker panel is combined with CRP for distinguishing bacterial from viral infections.
Prognostic value for sepsis severity (qSOFA ≥2) and adverse outcomes | At hospital admission (retrospective review of cases from September 1, 2021 to November 30, 2024)
  Assess the ability of the biomarker panel to predict clinical disease severity in patients with acute febrile illness, as measured by the qSOFA score.
Sensitivity, specificity, PPV, NPV, LR+/LR- for differentiating bacterial vs viral infection | At hospital admission (retrospective review of cases from September 1, 2021 to October 31, 2024)

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant-level clinical data and proteomic assay data generated from plasma samples will be shared.
Time Frame: Available after publication of primary results.
Access Criteria: Researchers with approved proposals and signed data-sharing agreements.